CLINICAL TRIAL: NCT00310271
Title: A Phase I Study Assessing Safety and Tolerability of a DNA Vaccine With a DNA Encoded Immunostimulator , Administered by Particle Mediated Epidermal Delivery Using the PowderMed ND10 Delivery System in HSV-2 Seronegative Healthy Volunteers
Brief Title: A Safety Study to Assess a DNA Vaccine Administered by Particle Mediated Delivery to the Skin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PowderMed (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PM HSD-001 P
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2008-11-21 (Estimated); Status verified 2008-11

CONDITIONS: HSV-2
Keywords: DNA vaccine, immunotherapy, HSV-2, PMED

INTERVENTIONS:
Biological: pPJV7630 with pPJV2012 administered by PMED

SUMMARY:
The purpose of this study is to evaluate how well the vaccine is tolerated at sites where administrations are given and any effects it may have on subjects' wellbeing. The study will also test the ability of vaccine to cause particular immune responses in the body.

DETAILED DESCRIPTION:
Herpes simplex virus type 2 (HSV-2) infection is a serious public health problem, with up to 20% of the US population infected. Following primary infection, HSV-2 establishes a latent infection that can lead to recurrent disease when the virus reactivates. Genital lesions are often experienced with viral recurrence and these can be uncomfortable and painful, resulting in significant anxiety and social distress. There are no commercial vaccines available for therapy of HSV-2 infection.The aim of a therapeutic vaccine would be to enhance such natural responses by boosting the appropriate cellular immune response to HSV-2 in those latently infected individuals who experience frequent and unwanted reactivations. The purpose of this study is to evaluate the safety and tolerability profile of a therapeutic DNA vaccine (pPJV7630) in combination with a DNA encoded immunostimulator (pPJV2012) when administered by Particle Mediated Epidermal Delivery (PMED)

ELIGIBILITY:
Otherwise healthy subjects with seronegative HSV-2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42
Dates: Start 2006-04; Study Completion 2006-12

PRIMARY OUTCOMES:
Safety, tolerability and reactogenicity of the investigational product as determined by AEs and evaluation of the site of vaccination at each visit.

SECONDARY OUTCOMES:
immunogenicity of vaccine post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Steven Komjathy, MD, Principal Investigator — PRA
Locations (1):
- CPC Phase I Unit, Lenexa, Kansas, United States